CLINICAL TRIAL: NCT04535596
Title: Comparison of Blood Flow Restriction Exercises With Conservative Exercises in Knee Osteoarthritis: A Randomized Controlled Single-Blind Study.
Brief Title: Blood Flow Restriction Exercises and Conservative Exercises in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, gizem ergezen, Gizem Ergezen, MSc, Physiotherapist, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10840098-722.02-E.34224
Record Dates: First submitted 2020-08-28; First posted 2020-09-02 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Osteoarthritis of Knee; Blood Flow Restriction Exercise; Resistance Training; Occlusion Training; Pain, Joint; Hypertrophy
MeSH Terms: conditions — Osteoarthritis, Knee; Arthralgia; Hypertrophy | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Exercises (Experimental): 12 week long strength training exercise with the higher loading (%70-80 of 1 Repetitive Maximum)
  Interventions: Other: Exercise
- Blood Flof Restriction Exercises (Experimental): 12 week long strength training exercise with the lower loading (%20-30 of 1 Repetitive Maximum) by using cuff around the thigh
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — 12 week long strength training exercises for knee

SUMMARY:
Knee osteoarthritis (OA) is a rheumatic disease that causes serious cartilage damage in the knee joint. Moderate physical activity can slow cartilage degeneration in moderate OA stages. Remarkable weakness and atrophy of the quadriceps and hamstrings is a common problem in patients with chronic osteoarthritis, but in arthritis, it may be difficult to achieve strength gains due to the pain caused by heavy load-resistant exercises. Exercising with these high loads may not be possible or may injure painful arthritic knees. For this reason, lately, blood flow restriction exercises have been directed to achieve the same gain by exercising with lower loads by restricting the blood flow with a cuff. We aimed to limit the blood flow in osteoarthritic knees and to provide strength gain and pain reduction provided by conventional exercises given routinely. Our hypothesis in this study is that exercises that blood flow restriction exercises will reduce pain and increase strength as well as conventional exercises.

DETAILED DESCRIPTION:
Knee osteoarthritis is a rheumatic disease that causes serious cartilage damage in the knee joint. Moderate physical activity can slow cartilage degeneration in moderate OA stages. Remarkable weakness and atrophy of the quadriceps and hamstrings is a common problem in patients with chronic osteoarthritis, but in arthritis, it may be difficult to achieve strength gains due to the pain caused by heavy load-resistant exercises. Exercising with these high loads may not be possible or may injure painful arthritic knees. For this reason, lately, blood flow restricting exercises have been directed to achieve the same gain by exercising with lower loads by restricting the blood flow with a cuff. We aimed to limit the blood flow in osteoarthritic knees and to provide strength gain and pain reduction provided by conventional exercises given routinely. Our hypothesis in this study is that exercises that limit blood flow will reduce pain and increase strength as well as conventional exercises. Forty patients diagnosed with knee osteoarthritis by X-ray will be included in the study. Grade II-III (high rate of exercise therapy) individuals according to the Kellgren Lawrence classification will be included. Patients diagnosed with orthopedics and traumatology will be randomly divided into two groups according to the order of entry through the door. Conventional Exercises that increase muscle strength, flexibility and reduce pain will be included in the first group. In the second group, the same exercises will be used, but during the application, a cuff will be placed on the thigh and the blood flow will be prevented by inflating, therefore, exercises with lower loads will be performed. Exercises will be practiced for 12 weeks and pre-exercise results will be compared within and between groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants between the ages of 45-70, diagnosed with knee osteoarthritis according to the criteria of the American College of Rheumatology.
* Participants who stated that the severity of knee pain to be evaluated with Visual Analog Pain Scale (VAS) is between 2-8
* Participants who are voluntaries for the study

Exclusion Criteria:

* Participants who have patellar subluxation or dislocation around the knee, who have other sources of knee pain such as bursae, fat pad and a history of knee surgery,
* Those who are in Grade 1 or 4 according to the Kellgren-Lawrence radiographic staging
* Those who have participated in leg weight exercise training in the last 6 months
* Participants who are under the high risk of venous thrombosis (lower extremity surgery, cardiovascular conditions including high blood pressure (> 140/90) in the past 6 months),
* Diabetes, pregnancy, unexplained chest pain or heart disease, fainting or dizziness during physical activity / exercise.
* If exercise is contraindicated

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 12 weeks
  Pain intensities which are assessed by visual analogue scale(VAS) divided 10 equal intervals. "0" means no pain and "10" means unbearable pain. Higher scores idicate worse pain intensity.
WOMAC score | 12 weeks
  score among patients with knee and/or hip osteoarthritis. The Index is self-administered, 24 question, 5-point Likert. Scores range from 0 to 96 for the total WOMAC where higher scores indicate worse function.

SECONDARY OUTCOMES:
high sensitive C-reactive protein (hs-CRP) | 12 weeks
  hs-CRP(high sensitive C-reactive protein) level
Physical Function | 12 weeks
  measured by 6 minute walking test
Physical Function | 12 weeks
  measured by sit-stand test
Physical Function | 12 weeks
  measured by timed up and go test,
Quadriceps muscle strength | 4 weeks
  peak isometric knee extensor torque measured by myometer.
Quadriceps cross sectional area | 12 weeks
  Measured by MRI
Circumference of thigh | 12 weeks
  measured in the same level of quadriceps before and after application.
Short Form-36 questionnaire | 12 weeks
  SF-36 quality of life form

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Ergezen, MSc, Principal Investigator — Medipol University; Mustafa Sahin, PhD, Principal Investigator — Medipol University; Candan Algun, PhD, Study Chair — Medipol University
Locations (1):
- Gizem Ergezen, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: starting 3 months after publication